CLINICAL TRIAL: NCT06239311
Title: A Phase 3, Randomised, 2-arm, Parallel-group, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Subcutaneous Methotrexate Versus Placebo in Moderate to Severe Atopic Dermatitis.
Brief Title: Efficacy and Safety of Methotrexate Versus Placebo in Adults With Atopic Dermatitis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC-MTX.18/AD; 2023-504443-13-00 (EU CTIS Number)
Record Dates: First submitted 2024-01-11; First posted 2024-02-02 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Moderate to Severe Atopic Dermatitis
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Active Comparator): Participants will receive 16 to 24 weekly subcutaneous injections of 20 mg . In case of intolerance of the 20 mg dose, a reduction to 15 mg per week is possible.
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Participants will receive 16 to 24 weekly subcutaneous injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Solution for injection in prefilled pen
  Arms: Methotrexate
Drug: Placebo — Solution for injection in prefilled pen
  Arms: Placebo

SUMMARY:
Atopic dermatitis is an ongoing condition that causes skin irritation, redness, and itchiness. Treatments are usually topical - applied to the skin (e.g., moisturisers or medicated creams) - but a wider variety of systemic treatments (that target the whole body) are needed for those whose condition does not improve with topical treatments. Methotrexate, a drug approved for similar conditions such as arthritis and psoriasis, has been shown to improve atopic dermatitis. This randomised, controlled clinical trial will investigate how effective.

ELIGIBILITY:
Inclusion Criteria:

* Woman of childbearing potential must have a negative pregnancy test at the Screening Visit and must agree to use highly effective methods of contraception while taking the investigational medicinal product (IMP) and for 6 months after the last IMP administration. Men must agree to use a condom during intercourse while taking the IMP and for 3 months after the last IMP administration. They must also agree to not donate sperm for the time period starting at the Screening Visit, throughout the entire trial period, and for at least 3 months after the last IMP administration.
* Diagnosis of atopic dermatitis (AD) at least 12 months prior to the Screening Visit, diagnosed as defined by the Hanifin and Rajka criteria for AD 4.
* Moderate to severe AD, defined as the following criteria at the Baseline Visit: Eczema Area and Severity Index (EASI) ≥ 16, Investigator Global Assessment (IGA) ≥ 3, Dermatology Life Quality Index (DLQI) ≥ 10
* Eligible for systemic treatment, ie, documented history (within 12 months prior to Baseline Visit) of inadequate response to treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI)s or documented systemic treatment for AD (such as cyclosporine (CYC), azathioprine and/or mycophenolate mofetil). Inadequate response to TCS or TCI is defined as failure to obtain or maintain a remission or a low activity disease (IGA ≥ 2) despite a daily treatment with a class 2 or class 3 TCS or TCI for 28 days (or the maximal authorised duration according to the Summary of Product Characteristics (SmPC))
* Treated with a stable dose of topical emollient, for at least 7 consecutive days prior to the Baseline Visit
* Chest X-ray without clinically relevant abnormalities performed within the last 6 months prior to the Baseline Visit
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Willing and able to comply with the protocol requirements for the duration of the trial
* Covered by health care insurance in accordance with local requirements

Exclusion Criteria:

* Pregnant or breast-feeding women, or planning to become pregnant, or to breastfeed during the trial
* Previously treated with MTX
* Presenting a known hypersensitivity to MTX or folic acid as well as to any of the excipients
* Presenting ulcers of the oral cavity and known active gastrointestinal ulcer disease
* Presenting with known blood dyscrasia (haemoglobin < 8.0 g/dL or white blood cell count < 4000/mm3 or platelet count < 100000/mm3)
* Presenting liver impairment and/or aspartate transaminase (AST) or alanine aminotransferase (ALT) > 2 times the upper limit of normal (ULN), or bilirubin > 5 mg/dL (85.5 μmol/L), or a positive result in the FibrotestTM at the Screening Visit
* Presenting drug or alcohol abuse within the last 12 months
* Presenting renal impairment (creatinine clearance less than 60 mL/min)
* Presenting serious, acute or chronic infections such as tuberculosis, hepatitis B or C, HIV positive, or other immunodeficiency syndromes

  1. A positive test result at Screening for hepatitis B surface antigen (HBsAg) and/or core antibodies (anti-HBc) excludes the patient from trial participation. Patients with positive surface antibodies (anti-HBs) and a history of hepatitis B virus (HBV) vaccination may be included.
  2. A positive test result at Screening for hepatitis C (positive hepatitis C virus (HCV) antibody test confirmed with positive hepatitis C RNA test) excludes the patient from trial participation, even if they have received appropriate and effective treatment, due to the risk of reactivation.
  3. If the interferon-gamma release assay shows a positive result at the Screening Visit the patient may only be included in the trial if the tuberculosis is latent and all of the following 3 conditions are true: (i) Chest X-ray does not show evidence suggestive of active tuberculosis. (ii) There are no clinical signs and symptoms of pulmonary and/or extra-pulmonary tuberculosis. (iii) Documented receipt of one of the following prophylactic treatment regimens: Oral daily isoniazid for 6 months or Oral daily rifampin for 4 months or Isoniazid and rifapentine weekly for 3 months. The IMP can only be administered to a participant with a positive test result in the interferon-gamma release assay (or an indeterminate result if only 1 test is done, or 2 indeterminate results if a second test is done after the first indeterminate test result) after the approval of a tuberculosis specialist.
* Presenting uncontrolled infection, hospitalisation due to uncontrolled infection or treatment with intravenous antibiotics for infection within 2 months prior to the Baseline Visit
* Presenting a history of malignancy, including solid tumours and haematologic malignancies, except non-melanoma skin cancer (epithelial cell carcinoma or basal cell carcinoma) and cervical carcinoma in situ that have been treated with no evidence of recurrence during the past 5 years
* Currently experiencing or having a history of other concomitant skin conditions that would interfere with evaluation of AD (eg. psoriasis, lupus erythematosus, eczema herpeticum)
* Treated with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before the Baseline
* Treated with TCS, calcineurin inhibitors or phosphodiesterase-4 inhibitors such as crisaborole within 1 week prior to the Baseline Visit
* Treated with oral corticosteroids, azathioprine, mycophenolate mofetil, CsA (Ciclosporin A) or any other systemic immunosuppressor / immunomodulator within 4 weeks before the Baseline Visit
* Treated by specific allergen immunotherapy started within 3 months before the Baseline Visit 17
* Treated with a monoclonal antibody (including but not limited to dupilumab or tralokinumab) within the last 3 months or 5 times the half-life of the respective monoclonal antibody (whichever is the longer period) or with any JAK (Janus kinase) inhibitors (including but not limited to ruxolitinib, baricitinib, tofacitinib, upadicitinib, or abrocitinib) within the last 4 weeks prior to the Baseline Visit
* Treated with any parenteral corticosteroid within 6 weeks prior to the Baseline Visit
* Treated with ultraviolet therapy within 4 weeks prior to the Baseline Visit
* Received a live (attenuated) vaccine within 4 weeks before the Baseline Visit or planning to be vaccinated with live vaccine during the trial. Please note: Since MTX may have an effect on the immune system, vaccination with live vaccines must not be performed during MTX administration
* Having a planned surgery during the trial
* Presenting a clinically significant medical disease that is uncontrolled despite treatment that, in the opinion of the Investigator, is likely to impact the ability to participate in the trial or to impact the trial efficacy or safety assessments
* Presenting any additional condition that, in the opinion of the Investigator, may interfere with the assessment or may put the participant at risk
* Protected by the law (adult under guardianship, or hospitalised in a public or private institution for a reason other than this trial, or incarcerated)
* Persons performing mandatory military service, persons deprived of liberty, persons who, due to a judicial decision, cannot take part in clinical trials, and persons, who due to their age, disability or state of health are reliant on care and for that reason accommodated in residential care institutions, that is accommodations providing an uninterrupted assistance for persons who necessitate such assistance, are in a situation of subordination or factual dependency and therefore may require specific protective measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) 75 response at Trial Week 16 Visit | Trial Week 16
  To demonstrate the superiority of subcutaneous (SC) methotrexate (MTX) versus placebo with respect to an improvement from baseline of at least 75% of the Eczema Area and Severity Index (EASI 75 response).
  The Eczema Area and Severity Index (EASI) is an investigator-assessed instrument for measuring the severity of clinical symptoms in atopic dermatitis (AD). The minimum EASI score is 0 (= normal) and the maximum EASI score is 72 (= very severe).

SECONDARY OUTCOMES:
Improvement from baseline of at least 50% in the Eczema Area and Severity Index (EASI 50 response) | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  The Eczema Area and Severity Index (EASI) is an investigator-assessed instrument for measuring the severity of clinical symptoms in atopic dermatitis (AD). The minimum EASI score is 0 (= normal) and the maximum EASI score is 72 (= very severe).
Improvement from baseline of at least 75% in the Eczema Area and Severity Index (EASI 75 response) | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 24
  The Eczema Area and Severity Index (EASI) is an investigator-assessed instrument for measuring the severity of clinical symptoms in AD. The minimum EASI score is 0 (= normal) and the maximum EASI score is 72 (= very severe).
Improvement from baseline of at least 90% in the Eczema Area and Severity Index (EASI 90 response) | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  The Eczema Area and Severity Index (EASI) is an investigator-assessed instrument for measuring the severity of clinical symptoms in atopic dermatitis (AD). The minimum EASI score is 0 (= normal) and the maximum EASI score is 72 (= very severe).
Change from baseline in the Eczema Area and Severity Index (EASI) score. | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  The Eczema Area and Severity Index (EASI) is an investigator-assessed instrument for measuring the severity of clinical symptoms in atopic dermatitis (AD). The minimum EASI score is 0 (= normal) and the maximum EASI score is 72 (= very severe).
Scoring Atopic Dermatitis (SCORAD) 50 response | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  Response is defined as an improvement from baseline of at least 50%.
  The Scoring Atopic Dermatitis (SCORAD) evaluates the extent and severity of eczema in atopic dermatitis (AD) based on affected body area and intensity of plaque characteristics.It comprises 3 areas: Area, Intensity and Subjective Symptoms. The final result range is between 0 (best result) and 103 (worst result).
Scoring Atopic Dermatitis (SCORAD) 75 response | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16,
  Response is defined as an improvement from baseline of at least 75%.
  The Scoring Atopic Dermatitis (SCORAD) evaluates the extent and severity of eczema in atopic dermatitis (AD) based on affected body area and intensity of plaque characteristics.It comprises 3 areas: Area, Intensity and Subjective Symptoms. The final result range is between 0 (best result) and 103 (worst result).
Change in Scoring Atopic Dermatitis (SCORAD) score from baseline | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  The Scoring Atopic Dermatitis (SCORAD) evaluates the extent and severity of eczema in atopic dermatitis (AD) based on affected body area and intensity of plaque characteristics.It comprises 3 areas: Area, Intensity and Subjective Symptoms. The final result range is between 0 (best result) and 103 (worst result).
Investigator Global Assessment (IGA) response | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16, Trial Week 24
  Investigator Global Assessment (IGA) response is defined as either an IGA score of 0 (clear) or 1 (almost clear) and a reduction of the score of at least 2 points.
  The IGA score is a 5-point scale with morphologic descriptors for each score to assess the severity of atopic dermatitis from 0 - Clear 4 - Severe.
Pruritus Numerical Rating Scale (NRS) response | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16, Trial Week 24
  The Pruritus Numerical Rating Scale (NRS) response is defined as a decrease of the worst daily Pruritus NRS score from baseline by at least 4 points in participants with an NRS of at least 4 points at baseline.
  The NRS is a single item designed to capture information on self-reported severity of worst itching each day on an 11-point scale from 0 ("no itch") to 10 ("worst itch imaginable").
Change from baseline in Pruritus Numerical Rating Scale (NRS) score | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  The Pruritus Numerical Rating Scale (NRS) is a single item designed to capture information on self-reported severity of worst itching each day on an 11-point scale from 0 (no itch) to 10 (worst itch imaginable).
Patient-oriented Eczema Measure (POEM) response | Trial Week 8, Trial Week 16
  Patient-oriented Eczema Measure (POEM) response is defined as reduction from baseline of at least 4 points.
  The POEM is a seven-item, patient-reported questionnaire assessing atopic dermatitis (AD)/eczema-specific symptoms over the last week; each item is scored 0 (no days) to 4 (every day) based on the number of days affected. The minimum POEM score is 0 (best result) and the maximum total POEM score is 28 (worst result).
Change from baseline in POEM score | Trial Week 8, Trial Week 16
  The POEM is a seven-item, patient-reported questionnaire assessing atopic dermatitis (AD)/eczema-specific symptoms over the last week; each item is scored 0 (no days) to 4 (every day) based on the number of days affected. The minimum POEM score is 0 (best result) and the maximum total POEM score is 28 (worst result).
Adverse events (AE), treatment-related AEs, serious adverse events (SAEs) and serious adverse reactions (SARs) | Trial Week 16, Trial Week 20, Trial Week 24, Trial Week 33
  For participants who have not reached EASI 50 by the Trial Week 16 Visit and do not enter the extension phase: Adverse events (AE), treatment-related AEs, serious adverse events (SAEs) occurring from the Screening Visit until Trial Week 16 Visit, and serious adverse reactions (SARs) occurring from start of the trial intervention until the Trial Week 20 Visit For participants who do reach EASI 50 by the Trial Week 16 Visit and do enter the extension phase: AEs, treatment-related AEs, SAEs occurring from the Screening Visit until End of Extension Visit (Trial Week 24), and SARs occurring from start of the trial intervention until the Follow-up Visit (Trial Week 33)
Dermatology Life Quality Index (DLQI) response | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  Dermatology Life Quality Index (DLQI) response is defined as reduction of at least 4 points in DLQI from baseline.
  The DLQI is a 10-item questionnaire assessing health-related quality of life over the last week in patients with dermatological symptoms, with each item scored for impact from not at all (0) to very much (3).
Change from baseline in Dermatology Life Quality Index (DLQI) score. | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  The Dermatology Life Quality Index (DLQI) is a 10-item questionnaire assessing health-related quality of life over the last week in patients with dermatological symptoms, with each item scored for impact from not at all (0) to very much (3).
Change from baseline in Scoring Atopic Dermatitis (SCORAD) sleep score | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  Scoring Atopic Dermatitis (SCORAD) sleep score is a subset of the SCORAD related to the subjective symptoms section (insomnia) sleeplessness will be evaluated by the participant (based on the quality of life in the past 3 days). A 10 cm visual analogue scale is used, with 0 for no symptom and 10 for most severe symptom.
Change from baseline in Work Productivity and Activity Impairment: General Health (WPAI:GH) | Trial Week 8, Trial Week 16
  The Work Productivity and Activity Impairment: General Health (WPAI:GH) questionnaire consists of 6 questions assessing the effect of AD (including physical and emotional problems or symptoms) on the participant's ability to work and to perform regular activities. The questions are computed according to specific calculation rules and have four scores. High scores indicate prolonged sick leave or impairment and decreased productivity.
Change from baseline in Hospital Anxiety and Depression (HADS) score and subscales | Trial Week 8, Trial Week 16
  Hospital Anxiety and Depression (HADS) is a fourteen-item scale with seven items each for anxiety and depression subscales. Each subscale can score between 0 (best result) and 21 (worst result) for either anxiety or depression.
Change from baseline in European Quality of Life (EuroQoL) Group 5 Dimension 5 Levels (EQ-5D-5L) | Trial Week 8, Trial Week 16
  The European Quality of Life (EuroQoL) Group 5 Dimension 5 Levels (EQ-5D-5L) consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises 5 dimensions, each dimension has 5 levels. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number ranging from 11111 (full health) to 55555 (worst health).
  The EQ VAS records the participant's self-rated health on a vertical visual analogue scale from 0 (The worst health you can imagine) to 100 (The best health you can imagine).
Change from baseline in Atopic Dermatitis Control Tool (ADCT) score | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  The Atopic Dermatitis Control Tool (ADCT) is a validated tool to evaluate the different dimensions of patient-perceived atopic dermatitis (AD) control. It consists of 6 questions, each scored from 0 to 4. The minimum total ADCT score is 0 (best result) and the maximum total ADCT score is 24 (worst result).
Eczema Area and Severity Index (EASI) 75 response at Trial Week 24 and the Follow-up Visit (Week 33) | Trial Week 24, Trial Week 33
  The Eczema Area and Severity Index (EASI) response in those participants who had an EASI 75 response at Trial Week 24 and did not need any systemic treatment for AD (relapse) until the Follow-up Visit.
  The EASI is an investigator-assessed instrument for measuring the severity of clinical symptoms in atopic dermatitis (AD). The minimum EASI score is 0 (= normal) and the maximum EASI score is 72 (= very severe).
Scoring Atopic Dermatitis (SCORAD) 90 response | Trial Week 4, Trial Week 8, Trial Week 12, Trial Week 16
  Response is defined as an improvement from baseline of at least 90%.
  The Scoring Atopic Dermatitis (SCORAD) evaluates the extent and severity of eczema in atopic dermatitis (AD) based on affected body area and intensity of plaque characteristics.It comprises 3 areas: Area, Intensity and Subjective Symptoms. The final result range is between 0 (best result) and 103 (worst result).

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Nosbaum, MD PhD, Principal Investigator — Université Lyon 1 / INSERM U1111 - CIRI / Hospices Civils de Lyon
Locations (30):
- Czechia (8):
  - MU Dr. Petr Arenberger, DrSc. MBA, Prague, Praha 1
  - Synexus Czech s.r.o., Prague, Praha 2
  - Praglandia s.r.o., Prague, Praha 5
  - AGE Centrum s.r.o., Olomouc
  - CCR Ostrava s.r.o,, Ostrava
  - CCR Czech Pardubice a.s., Pardubice
  - Clintrial s.r.o., Prague
  - Dermatology clinic MUDr. Blanka Havlickova, Prague
- France (4):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Saint Andre, Bordeaux
  - Centre Hospitalier universitaire (CHU) de Clermont Ferrand Hopital d'Estaing, Clermont-Ferrand
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
- Italy (6):
  - Ospedale San Donato di Arezzo, Arezzo
  - Azienda Ospedaliera Universitaria di Ferrara Arcispedale Sant' Anna, Ferrara
  - Ospedale Piero Palagi, Florence
  - Universita degli Studi della Campania "Luigi Vanvitelli" - Azienda Ospedaliera Universitaria, Naples
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Ospedaliero Universitaria Pisana (AOUP), Pisa
- Poland (12):
  - Synexus Polska Sp. z o.o. in Czestochowa, Częstochowa
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Angelius Badania Kliniczne, Katowice
  - Synexus Polska Sp. z. o.o. Oddzial W Lodzi, Lodz
  - LUXDERM Specjalistyczny Gabinet Dermatologiczny Prof. dr hab. n. med. Dorota Krasowska, Lublin
  - Klinika Zdybski, Lublin
  - Twoja Klinika, Mikołów
  - Synexus Polska Sp z o.o. Oddzial W Poznaniu, Poznan
  - Laser Clinic, Szczecin
  - Synexus Polska Sp. Z o.o. Odział w Warszawie, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw